CLINICAL TRIAL: NCT02087241
Title: A Phase II Study of AZD1775 Plus Pemetrexed and Carboplatin Followed by a Randomised Comparison of Pemetrexed and Carboplatin With or Without AZD1775 in Patients With Previously Untreated Stage IV Non-Squamous Non-Small-Cell Lung Cancer
Brief Title: Ph II Trial of Carboplatin and Pemetrexed With or Without AZD1775 for Untreated Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The sponsor decided to terminate the study.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D6011C00002
Record Dates: First submitted 2014-03-06; First posted 2014-03-14 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Previously Untreated Stage IV Non-Squamous Non Small Cell Lung Cancer
Keywords: Stage IV Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — adavosertib; Pemetrexed; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZD1775 + carboplatin + pemetrexed (Experimental): Randomised: AZD1775 + pemetrexed + carboplatin followed by maintenance AZD1775 + pemetrexed versus pemetrexed and carboplatin followed by maintenance pemetrexed.
  Interventions: Drug: AZD1775; Drug: pemetrexed; Drug: carboplatin
- Placebo + carboplatin + pemetrexed (Experimental): Randomised: AZD1775 + pemetrexed + carboplatin followed by maintenance AZD1775 + pemetrexed versus pemetrexed and carboplatin followed by maintenance pemetrexed.
  Interventions: Drug: AZD1775 Matching Placebo; Drug: pemetrexed; Drug: carboplatin

INTERVENTIONS:
Drug: AZD1775 — AZD1775 is a highly selective, adenosine-triphosphate (ATP) competitive, small molecule inhibitor of the WEE 1 kinase that sensitizes tumor cells to cytotoxic agents and is being developed for the treatment of advanced solid tumors and p53 pathway deficient malignancies
  Other Names: MK-1775
  Arms: AZD1775 + carboplatin + pemetrexed
Drug: AZD1775 Matching Placebo — AZD1775 is a highly selective, adenosine-triphosphate (ATP) competitive, small molecule inhibitor of the WEE 1 kinase that sensitizes tumor cells to cytotoxic agents and is being developed for the treatment of advanced solid tumors and p53 pathway deficient malignancies
  Arms: Placebo + carboplatin + pemetrexed
Drug: pemetrexed — This drug is a part of a general group of chemotherapy drugs called anti-metabolites. It prevents cells from using folate to make DNA and RNA. Because cancer cells need these substances to make new cells, this drug helps to stop the growth of cancer cells.
Drug: carboplatin — This drug is a platinum chemotherapy drug that acts like an alkylating agent. It stops the growth of cancer cells, causing the cells to die.

SUMMARY:
The aim of this study is to combine AZD1775 with standard front-line chemotherapy in subjects with advanced NSCLC.

DETAILED DESCRIPTION:
This is a randomised, phase II trial comparing AZD1775 plus pemetrexed and carboplatin followed by maintenance AZD1775 and pemetrexed versus pemetrexed and carboplatin followed by maintenance pemetrexed in patients with previously untreated metastatic non-squamous NSCLC with TP53 mutations. The primary endpoint of the trial is assessment of progression-free survival (PFS).

ELIGIBILITY:
Inclusion Criteria

* Provision of informed consent prior to any study specific procedures
* Histologic or cytologic diagnosis of advanced NSCLC, Recurrent or Stage IV disease (according to American Joint Committee on Cancer (AJCC) staging system, v7.0).
* No prior chemotherapy for locally advanced or metastatic disease
* Subjects with a known EGFR mutation must have received previous treatment with an EGFR tyrosine kinase inhibitor; and subjects with a known ALK translocation must have received previous treatment with an ALK inhibitor.
* No prior radiation therapy to the whole pelvis or to ≥25% of the total bone marrow area.
* At least one measurable lesion according to Response Evaluation Criteria in Solid Tumours (RECIST) v1.1
* Mandatory availability of tumour tissue (archival or fresh if archival is not available) for TP53 determination.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0 or 1.
* Absolute neutrophil count (ANC) ≥1500/μL
* Hemoglobin (Hgb) ≥10 g/dL
* Platelets ≥100,000/μL
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST), ≤3.0 x the upper limit of normal (ULN); 5 x ULN if known hepatic metastases
* Total bilirubin ≤1.5 x ULN, unless secondary to Gilbert's disease
* Serum creatinine ≤1.5 x ULN and a calculate creatinine clearance (CrCl) ≥45 mL/min by the Cockcroft-Gault method
* Ability to swallow oral medication
* Fertile male subjects willing to use at least one medically acceptable form of birth control for the duration of the study and for 2 weeks after treatment stops
* Female subjects who are not of childbearing potential and fertile female subjects of childbearing potential who agree to use adequate contraceptive measures who are not breastfeeding, and who have a negative serum or urine pregnancy test within 72 hours prior to start of study treatment
* Predicted life expectancy ≥12 weeks
* Must be ≥18 years of age
* Willingness and ability to comply with study and follow-up procedures
* Ability to understand the nature of this trial and give written informed consent Exclusion criteria
* Use of a study drug ≤21 days or 5 half-lives (whichever is shorter) prior to the first dose of AZD1775
* Major surgical procedures ≤28 days of beginning AZD1775, or minor surgical procedures ≤7 days
* Known central nervous system (CNS) disease
* Subject has had prescription or non-prescription drugs or other products (i.e. grapefruit juice) known to be sensitive CYP3A4 substrates
* Any known hypersensitivity or contraindication to the components of study treatment
* Any of the following cardiac diseases currently or within the last 6 months as defined by New York Heart Association ([NYHA] Appendix G) ≥ Class 2
* Corrected QT interval (QTc) >470 msec (as calculated by Fridericia correction formula) at study entry or congenital long QT syndrome.
* Pregnant or lactating
* Any serious, active underlying medical condition that would impair the ability of the subjects to receive study treatment
* Unable or unwilling to take folic acid or vitamin B12
* Presence of other active cancers, or history of treatment for invasive cancer ≤3 years
* Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R Spigel, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (8):
- United States (8):
  - Research Site, Englewood, Colorado
  - Research Site, Fort Myers, Florida
  - Research Site, Orlando, Florida
  - Research Site, Peoria, Illinois
  - Research Site, Fort Wayne, Indiana
  - Research Site, Wichita, Kansas
  - Research Site, Cincinnati, Ohio
  - Research Site, Nashville, Tennessee

REFERENCES:
- [Derived] Johnson ML, Dakhil SR, Beck JT, Sadiq A, Menon S, Mugundu GM, Chmielecki J, Spigel DR. Two Phase II Trials of Adavosertib, a Wee1 Inhibitor with Docetaxel or Carboplatin plus Pemetrexed in Non-small-cell Lung Cancer. Target Oncol. 2025 Nov;20(6):967-978. doi: 10.1007/s11523-025-01177-x. Epub 2025 Nov 10. PMID 41212474

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 16 clinical sites in the United States. A total of 14 subjects were enrolled between March 19, 2014 and April 16, 2015.
Pre-assignment Details: 22 subjects were consented; 3 subjects failed screening. The study was terminated prior to the start of screening for 5 participants. 14 participants were treated with AZD1775. The study was terminated early by the sponsor. Part 2 was not done. The 14 participants were enrolled in 4 Cohorts, designated Cohorts 1, 2, 3, and A.
Groups:
- Cohort 1: AZD1775 225 mg bid. 5 doses over 3 days (Days 1, 2, and 3 of a 21- Day Cycle)/Pemetrexed 500 mg/Carboplatin AUC 6
- Cohort 2: AZD1775 225 mg bid. 5 doses over 3 days (Days 3, 4, and 5 of a 21-Day Cycle)/Pemetrexed 500 mg/Carboplatin AUC 6.
- Cohort 3: AZD1775 175 mg bid. 5 doses over 3 days (Days 3, 4, and 5 of a 21-Day Cycle)/Pemetrexed 500 mg/Carboplatin AUC 6
- Cohort A: AZD1775 125 mg bid. 5 doses over 3 days (Days 1, 2, and 3 of a 21- Day Cycle)/Pemetrexed 400 mg/Carboplatin AUC 5
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort A
Started | 3 | 3 | 1 | 7
Completed | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 1 | 7
Not completed — Death | 2 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1
Not completed — Progressive Disease | 0 | 0 | 0 | 1
Not completed — Study Terminated by Sponsor | 0 | 2 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort A | Total
Number analyzed (Participants) | 3 | 3 | 1 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.3 (6.03) | 59.0 (4.36) | 81.0 (0) | 62.6 (9.41) | 63.7 (8.88)
Age, Continuous [Median (Full Range); unit: Years] | 66.0 [59 to 71] | 61.0 [54 to 62] | 81.0 [81.0 to 81.0] | 64.0 [46 to 73] | 63.0 [46 to 81]
Age, Customized [Number; unit: Participants]
  < 65 | 1 | 3 | 0 | 4 | 8
  >= 65 | 2 | 0 | 1 | 3 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 0 | 3 | 8
  Male | 1 | 0 | 1 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 3 | 2 | 1 | 7 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1
  White | 3 | 3 | 1 | 6 | 13
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  United States | 3 | 3 | 1 | 7 | 14
Tobacco Use [Number; unit: Participants]
  Smoker | 3 | 3 | 1 | 7 | 14
  Non-Smoker | 0 | 0 | 0 | 0 | 0
ECOG Performance Status [Number; unit: Participants] — The Eastern Cooperative Oncology Group (ECOG) scores are defined as follows: 0 = Asymptomatic (Fully active, able to carry on all predisease activities without restriction); 1 = Symptomatic but completely ambulatory (Restricted in physically strenuous activity and able to carry out work of a light or sedentary nature); 2 = Symptomatic, <50% in bed during the day; 3 = Symptomatic, >50% in bed, but not bedbound; 4 = Bedbound (Completely disabled. Cannot carry on any self-care; 5 = Dead
  Participants
    ECOG Performance Status = 0 | 1 | 1 | 1 | 3 | 6
    ECOG Performance Status = 1 | 2 | 2 | 0 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression free survival is defined as the time from randomisation until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the subject withdraws from randomised therapy or receives another anti-cancer therapy prior to progression.
Time Frame: 6 months
Population: Progression-Free Survival data were not collected.
Groups:
- Cohort 1: AZD1775 225 mg bid. 5 doses over 3 days (Days 1, 2, and 3 of a 21-Day Cycle)/Pemetrexed 500 mg/Carboplatin AUC 6.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort A
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Assess the Objective Response Rates in Each Arm
Description: The objective response rate is defined as the number of the subjects with a confirmed best overall response of CR or PR divided by the number of subjects in the Full Analysis Set (FAS) for whom measureable disease is present at baseline
Time Frame: Up to a maximum of 4 treatment cycles (treatment cycles will be repeated every 21 days)
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Groups:
- Cohort 2: AZD1775 225 mg bid. 5 doses over 3 days (Days 3, 4, and 5 of a 21- Day Cycle)/Pemetrexed 500 mg/Carboplatin AUC 6
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort A
Number analyzed (Participants) | 3 | 3 | 1 | 7
Percentage of Participants | 66.7 [13.54 to 98.30] | 33.3 [1.70 to 86.46] | 0 [0 to 0] | 14.3 [0.85 to 58.18]

3. Secondary Outcome: Assess the Disease Control Rate in Each Treatment Arm
Description: the disease control rate is defined as the percentage of FAS subjects with a best overall response of CR, PR or SD).
Time Frame: Up to a maximum of 4 treatment cycles (treatment cycles will be repeated every 21 days)
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Groups:
- Cohort A: AZD1775 125 mg bid. 5 doses over 3 days (Days 1, 2, and 3 of a 21-Day cycle)/Pemetrexed 400 mg/Carboplatin AUC 5
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort A
Number analyzed (Participants) | 3 | 3 | 1 | 7
Percentage of Participants | 66.7 [13.54 to 98.30] | 66.7 [13.54 to 98.30] | 0 [0 to 0] | 85.7 [60.70 to 100]

4. Secondary Outcome: Assess the Duration of Response in Each Treatment Arm
Description: Duration of response is defined as the time from the date of first documented response until the date of documented progression or any cause death.
Time Frame: Up to a maximum of 4 treatment cycles (treatment cycles will be repeated every 21 days)
Population: Duration of response data were not collected.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort A
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Assess Overall Survival in Each Treatment Arm
Description: Overall survival is defined as the time from the date of randomization until death due to any cause.
Time Frame: Up to a maximum of 4 treatment cycles (treatment cycles will be repeated every 21 days)
Population: Overall Survival (OS) data were not collected.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort A
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year, 3 months
Description: Adverse event data were collected from the time the first patient received the first dose of investigational drug on March 19, 2014 until the study was closed on June 1, 2015.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort A
Serious Adverse Events (participants affected / at risk) | 1/3 | 3/3 | 1/1 | 3/7
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 1/1 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=3) | Cohort 3 (N=1) | Cohort A (N=7)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MUCOSAL INFLAMMATION (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=3) | Cohort 3 (N=1) | Cohort A (N=7)
ANAEMIA (Blood and lymphatic system disorders) | 2 (2) | 1 (5) | 1 (1) | 2 (3)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 1 (4) | 0 (0) | 3 (5)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 (3) | 2 (8) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0/0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 2 (4) | 2 (2) | 1 (1) | 1 (1)
DUODENITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
GLOSSITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 3 (3) | 1 (4) | 1 (1) | 2 (6)
OESOPHAGITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 3 (5) | 0 (0) | 1 (1) | 2 (2)
ASTHENIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CHEST PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHILLS (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (5)
MUCOSAL INFLAMMATION (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
PERIPHERAL SWELLING (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OESOPHAGEAL CANDIDIASIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ORAL CANDIDIASIS (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0/1 (0) | 0 (0) | 1 (1)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 2 (3) | 1 (4) | 0 (0) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 1 (2) | 2 (9) | 0 (0) | 0 (0)
TROPONIN INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
WEIGHT DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 (0) | 1 (6) | 0 (0) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 4 (4)
DEHYDRATION (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (3)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (4) | 1 (1) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (8) | 0 (0) | 0 (0)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
SEBORRHOEIC KERATOSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ANXIETY (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
INSOMNIA (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHROMATURIA (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DYSURIA (Renal and urinary disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
VULVOVAGINAL BURNING SENSATION (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
PHLEBITIS SUPERFICIAL (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated on June 1, 2015 by the sponsor. The Primary Outcome Measure (Progression Free Survival) was not assessed and the randomised portion of the study was not done.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No